CLINICAL TRIAL: NCT05888675
Title: Randomized Clinical Trial:Clinical Study of Weifuchun Treatment on Gastric Cancer
Brief Title: Clinical Study of Weifuchun Treatment on Gastric Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: ShuGuang Hospital (Other)
Responsible Party: Principal Investigator, Mingyu Sun, Clinical Professor, ShuGuang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 42507214-10
Record Dates: First submitted 2023-04-28; First posted 2023-06-05 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Gastric Cancer (Diagnosis)
Keywords: Weifu Chun; Gastric Cancer; Clinical Efficacy; randomized clinical trial; mechanism
MeSH Terms: conditions — Stomach Neoplasms; Disease | interventions — weifuchun

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical Study of Weifuchun Treatment on Gastric Cancer (Other): 72 patients with gastric cancer were randomly divided into a treatment group of 36 cases and a control group of 36 cases. The treatment group received combination chemotherapy with Weifuchun tablets, while the control group received monotherapy chemotherapy.
  Interventions: Drug: Weifuchun

INTERVENTIONS:
Drug: Weifuchun — The treatment group#Weifuchun group#was given Weifuchun tablets, 4 tablets each time, 3 times a day, and 1 hour after meals. The control group(chemotherapy group)#Chemotherapy regimen was based on the Chinese Clinical Oncology Association Guidelines for the Diagnosis and Treatment of Gastric Cancer (2018), including oxaliplatin +5-FU/CF, SOX regimen, XELOX regimen, and Ticeo monotherapy regimen.

SUMMARY:
Research purpose To elucidate the effect mechanism and clinical effective of weifuchun in the prevention and treatment of gastric cancer. From genes related to cell differentiation, proliferation, apoptosis, tumor invasion and metastasis, genes related to immune inflammation and immune escape and other possible aspects to elucidate the effective and mechanism of weifuchun's treatment on gastric cancer.

DETAILED DESCRIPTION:
Weifuchun Treatment and mechanism on Gastric Cancer. Main Responsibility Person: Mingyu Sun research center#Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine Trial Objective#Observe the clinical efficacy and mechanism of Weifuchun in the treatment gastric cancer Therapeutic Schedule#In this study, 72 patients with gastric cancer who received chemotherapy in the Department of Gastrointestinal Surgery and Oncology, Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine were recruited and divided into groups according to random number table method, namely, 36 patients in the Weifichun combined chemotherapy group and 36 patients in the chemotherapy group alone. Weichun group was treated with 24 weeks of Chinese patent medicine Weichun tablet at the same time of chemotherapy. The physical status score, TCM syndrome score, quality of life score, bone marrow suppression and tumor index of the two groups before and 24 weeks after treatment were observed and compared.Fecal samples of the above patients before and after the entry and exit groups were collected, screened and submitted for examination. Finally, 15 cases were submitted for examination in the Weifichun combined chemotherapy group and chemotherapy group alone, and 10 cases were submitted for examination in the healthy volunteers. Miseq platform was used to conduct high-throughput sequencing and analysis of 16S ribosomal RNA of intestinal flora, fecal quality assessment of intestinal flora tested was conducted, α diversity and β diversity were analyzed, and the flora structure, including the level of taxonomy, family, genus, etc., were compared to analyze the differences in each group, and elucidate the possible mechanism of action of Weichun in the treatment of gastric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should be aged between 18 and 70 years old (including 18 and 70 years old) and their gender is not limited.
2. Pathological diagnosis of gastric malignant tumor;
3. The pathological types were adenocarcinoma, tubular adenocarcinoma, mucous adenocarcinoma and sig-ring cell carcinoma (including adenocarcinoma and some sig-ring cell carcinoma);
4. Patients were willing to receive chemotherapy (oxaliplatin +5-FU/CF, SOX regimen, XELOX regimen, or Ticeo monotherapy regimen).
5. The patient was willing to receive weifunchun treatment.

Exclusion Criteria:

1. Incomplete pathological diagnostic data;
2. Patients with severe heart, lung, liver, kidney (creatinine greater than the upper limit of the normal range), endocrine, hematopoietic system or psychiatric diseases were considered not suitable for the study group;
3. Pregnant or lactating women, as well as pregnant persons who may not have taken effective contraceptive measures;
4. People who are allergic (allergic to two or more kinds of food, drugs, etc.) or are allergic to known ingredients of the medicine;
5. Patients with other medical conditions that interfere with the trial and are deemed unsuitable for inclusion in the trial by the investigator;
6. Patients enrolled in other clinical trials within the last 1 month.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | the patients' were included into the clinical trials and up to 24 weeks treatment.
  To observe the effects of treatment group and control group on OS in patients with advanced gastric cancer, and evaluate whether there is statistical difference in OS between the two groups.From date of randomization until the date of death from any cause, whichever came first, assessed up to 24 months.

SECONDARY OUTCOMES:
Progression-free survival | the patients' were included into the clinical trials and up to 24 weeks treatment.
  The time between the first treatment and tumor progression or death.From date of randomization until the date of first documented progression, whichever came first, assessed up to 24 months. To observe the effects of treatment group and control group on PFS in patients with advanced gastric cancer, and evaluate whether there is a statistical difference in PFS between the two groups.
EORTC QLQ-C30 | the patients' were included into the clinical trials and up to 24 weeks treatment.
  The quality of life score is based on the EuroPean organization for Research and Treatment (EORTC) Quality of Life Scale (QLQ-C30 v3.0), which records changes in quality of life before and after treatment and compares them. Linear transformation of statistical results was performed to obtain standardized scores (0~100 points), so that scores in various fields could be compared with each other, and the problem of reverse entries could be solved at the same time. The higher the score of symptom field obtained by each subscale, the worse the quality of life condition. The higher the scores in the areas of function and general health, the better the patient's quality of life. Analyze whether there was a statistical difference between the two groups.
Clinical symptoms | the patients' were included into the clinical trials and up to 24 weeks treatment.
  According to the scoring criteria of the Guidelines for Clinical Research of New Chinese Medicines (2002), the symptoms of patients after treatment were determined. The improvement of patients' overall symptoms was evaluated by Nimodipine method, and the efficacy index after treatment = (total score before treatment - total score after treatment)/total score before treatment *100%.
Tumor markers | the patients' were included into the clinical trials and up to 24 weeks treatment.
  Detect the biomarkers (CA72-4, CEA, CA19-9, CA242, CA50, CA125) of two groups of patients before and after treatment to determine whether there is a statistical difference between the two groups before and after treatment.
Immune function | the patients' were included into the clinical trials and up to 24 weeks treatment.
  T cell subsets of the two groups were detected before and after treatment to determine whether there was a statistical difference between the two groups before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mingyu Sun, doctor, Principal Investigator — Ethics Committee of Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine

IPD SHARING:
Plan to Share IPD: Undecided